CLINICAL TRIAL: NCT01481675
Title: Resolution of Diabetes and Hormonal Changes Following Biliopancreatic Diversion Long Limbs and Laparoscopic Sleeve Gastrectomy. A Comparative Prospective Study.
Brief Title: Diabetes Resolution and Hormone Changes After BPDLL and LSG
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Theodore K. Alexandrides, Professor of Medicine, Head of Endocrine Division, University of Patras
Other Study IDs: BPDLSG002; BPDLL vs LSG (Other: University Hospital of Patras)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus
Keywords: biliopancreatic diversion; sleeve gastrectomy; diabetes mellitus; weight loss; ghrelin; PYY; GLP-1
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BPDLL group: Patients subjected to the Biliopancreatic Diversion Long Limbs surgical operation will undergo an oral glucose tolerance preoperatively and 12 months after the operation
- LSG group: Patients subjected to laparoscopic sleeve gastrectomy will undergo an oral glucose tolerance test preoperatively and 12 months postoperatively

SUMMARY:
To evaluate and compare prospectively the effects of Biliopancreatic Diversion Long Limb (BPDLL) and Laparoscopic Sleeve Gastrectomy (LSG) on resolution of diabetes mellitus type 2.

DETAILED DESCRIPTION:
Twelve patients with diabetes mellitus type 2 (DM 2) and body mass index (BMI)> 50kg/m2) will undergo BPDLL and 12 twelve patients with DM 2 and BMI 40-50 kg/m2 will undergo LSG. The patients will be evaluated before and 1, 3 and 12 months after surgery with an oral glucose tolerance test. The investigators aim to investigate the effects of surgery on diabetes resolution, hypertension, dyslipidemia, and also on fasting, and glucose-stimulated insulin, glucagon, ghrelin, peptide-YY and glucagon-like peptide-1 (GLP-1) responses during during an oral glucose tolerance test (OGTT). Resolution of diabetes mellitus will be evaluated according to the criteria of American Diabetes Association with an OGTT. The effects on appetite and satiety will be also evaluated with the use of visual analog scores.

ELIGIBILITY:
Inclusion Criteria:

* BMI>50kg/m2 to undergo BPDLL
* BMI 40-50kg/m2 to undergo LSG
* Diabetes mellitus type 2

Exclusion Criteria:

* Chronic medical illness
* Psychiatric illness
* Substance abuse
* Previous gastrointestinal surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twelve patients with diabetes mellitus type 2 and BMI> 50kg/m2 will undergo BPDLL and 12 patients with diabetes mellitus type 2 and BMI 40-50kg/m2 will undergo LSG
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Diabetes resolution at 12 months after surgery | 12 months after surgery

SECONDARY OUTCOMES:
Weight loss at 12 months after surgery | 12 months after surgery
Changes of GLP-1 response to glucose | 12 months after surgery
Changes in ghrelin levels | 12 months after surgery
Changes in PYY response to glucose | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Alexandrides, Professor, Principal Investigator — University of Patras; Fotis Kalfarentzos, Professor, Study Director — University of Patras
Locations (1):
- University Hospital of Patras, Rio, Achaia, Greece